CLINICAL TRIAL: NCT05127356
Title: Diagnostic Accuracy of DIAGNOdent Compared to ICDAS II in Detection of Incipient White Spot Lesions: An In-vivo Evaluation
Brief Title: Diagnostic Accuracy of DIAGNOdent Compared to ICDAS II
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Omar Osama Shaalan, Lecturer, Conservative Dentistry Department, Faculty of Dentistry, Cairo University
Other Study IDs: Diagnodent
Record Dates: First submitted 2021-11-05; First posted 2021-11-19 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Caries; Initial

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Laser fluorescence: DIAGNOdent is a laser fluorescence device that detects and quantify stages of development of incipient carious lesions
  0-4 healthy tooth structure; 5-10 Outer half enamel caries; 11-20 Inner half enamel caries; 21+ Dentin caries
  Interventions: Device: DIAGNOdent
- Visual examination: ICDAS II
  Code 0: Sound tooth surface; Code 1: First visual change in enamel; Code 2:Distinct visual change in enamel when viewed wet; Code 3: Localized enamel breakdown due to caries with no visible dentin; Code 4: Underlying dark shadow from dentin with or without localized enamel breakdown; Code 5: Distinct cavity with visible dentin; Code 6: Extensive distinct cavity with visible dentin.
  Interventions: Diagnostic Test: ICDAS II

INTERVENTIONS:
Device: DIAGNOdent — Laser fluorescence device
  Groups: Laser fluorescence
Diagnostic Test: ICDAS II — International Caries Detection and Assessment System (ICDAS II)
  Groups: Visual examination

SUMMARY:
There is a paradigm shift in conservative dentistry by substituting the surgical model with the medical model of treatment. Early detection of initial carious lesions will aid in clinical decision making during management ; either no care advised, preventive care advised or operative care advised. According to recent systematic reviews meticulous visual examination using ICDAS II presented a substantial level of reproducibility and accuracy for assessment of carious lesions and was considered the reference for clinical visual assessment . However, visual examination is subjective and is highly dependent on the dentist's skills and experience, with high specificity and low sensitivity. New devices have been developed to detect and quantify incipient demineralization. Besides visual detection systems, laser fluorescence assessment can be considered a suitable method. In vitro data suggested that the visual examination and fluorescence method have similar accuracy to detect initial carious lesions.

DETAILED DESCRIPTION:
This study will be conducted to evaluate the diagnostic accuracy of laser fluorescence device (DIAGNOdent) compared to to visual examination (ICDAS II) in detection of incipient carious lesions for decision making during caries management

ELIGIBILITY:
Inclusion Criteria:

* Non cavitated white spot lesions.
* Patient compliance

Exclusion Criteria:

* Cavitated lesions.
* Medically compromised patients.
* Enrollment in another clinical trials.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients with non cavitated incipient carious white spot lesions
Sampling Method: Non-Probability Sample
Enrollment: 193 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-05-05 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy | Immediate (cross-sectional)
  Assessing the validity of both methods in detecting initial carious lesions in terms of sensitivity and specificity.

CONTACTS AND LOCATIONS:
Overall Officials: Omar O Shaalan, PhD, Principal Investigator — Lecturer, Conservative Dentistry Department, Faculty of Dentistry, Cairo University
Locations (1):
- Faculty of Dentistry, Cairo University, Cairo, El Manial, Egypt

IPD SHARING:
Plan to Share IPD: No